CLINICAL TRIAL: NCT02093104
Title: Utilizing Intraprocedural Flow and Perfusion Dynamics as a Predictor of Response in Patients With Unresectable Hepatocellular Carcinoma Undergoing Chemoembolization and Radioembolization (Y90) "Liver Embolization Perfusion TACE Study (Version 1.0) EPTS 2013-1.0"
Brief Title: TACE Study-Liver Embolization Perfusion (VGH Radiology LIU)
Acronym: TACE
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Dave Liu, Principal Investigator, University of British Columbia
Other Study IDs: H12-03704; SIEMENS Canada/USA (Other: UBC CREB)
Record Dates: First submitted 2014-03-10; First posted 2014-03-20 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Unresectable Hepatocellular Carcinoma; Undergoing Chemoembolization and Radioembolization
Keywords: unresectable hepatocellular carcinoma; (undergoing chemoembolization and radioembolization)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to evaluate the quantitative information of utilizing C-arm systems in liver tumor care in hopes this potential clinical combination of imaging could aid in diagnosis and evaluation of tumor therapy.

DETAILED DESCRIPTION:
Blood flow imaging for liver tumors is normally carried out using clinical Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) systems prior to going to the cath lab. This study aims to determine if measuring flow using a C-arm system and/or CT perfusion can be used to improve diagnosis and evaluation of liver tumors.

The major difference between C-arm CT systems and clinical CT systems is the difference in imaging speed. We have developed a new approach that should allow us to overcome this speed limitation. The major difference between conventional CT versus CT perfusion is the obtaining of an extra series of images. CT perfusion results in an increase in the amount of radiation exposure during the CT scan that measures the blood flow of the targeted tumor; however, CT perfusion is much faster than conventional CT.

Prospective participants are being invited to the study because part of the treatment towards the tumour therapy involves obtaining an angiogram.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological diagnosis or meet the AASLD criteria for diagnosis of hepatocellular carcinoma (HCC) and at least one uni-dimensional lesion measurable according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria by CT-scan
2. OR radiologic evidence of liver metastatic disease
3. Amenable to embolization or ablation as adjuvant, neoadjuvant or definitive (curative or palliative) therapy.
4. Adult > 19 years old and estimated life expectancy over 3 months
5. Eastern Cooperative Oncology Group (ECOG) performance status under or equals 1
6. Adequate haematological function: Hb over or equals 9g/100mL, absolute neutrophil count over or equals 1 500/mm3, platelet count over or equals 50 000/mm3
7. Adequate renal function; serum creatinine under 150μmol/L
8. Bilirubin under or equals 50 µmol/L, Aspartate aminotransferase (AST) or ALT uner or equals 5 x upper limit of normal (ULN), international normalized ratio (INR) under or equals 1.5
9. Liver cirrhosis Child Pugh A - B7
10. Ability to provide written informed consent

Exclusion Criteria:

1. Advanced liver disease with Child-Pugh score over 7 or active gastrointestinal bleeding or encephalopathy or ascites refractory to diuretic therapy
2. Women who are pregnant or breast feeding
3. Allergy to contrast media
4. Contraindication to hepatic artery catheterisation, such as severe peripheral vascular disease precluding catheterisation OR contraindication to locally curative ablation due to size, location or shape.
5. Psychiatric or other disorder likely to impact on informed consent
6. Patient unable and/or unwilling to comply with treatment and study instructions

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with unresectable hepatocellular carcinoma undergoing chemoembolization and radioembolization
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Liver Tumour Perfusion using CT & C-arm systems in 40 patients at VGH over a 3 month period | 3 months
  The purpose of this protocol is to study the potential predictive and prognostic value of tumor perfusion assessment utilizing computed tomography and C-arm systems in the treatment of liver tumors.
  Observational nature of study; post hoc analysis precludes determination of primary endpoint.
  3 month follow-up CT scans as per protocol involving standard of care 4 phase CT scan in addition to perfusion CT
  Utilizing intraprocedural flow and perfusion dynamics as a predictor of response in 40 patients with unresectable hepatocellular carcinoma undergoing intraprocedural flow and perfusion dynamics as a predictor of response in chemoembolization and radioembolization (Y90)

CONTACTS AND LOCATIONS:
Overall Officials: David MT Liu, MD, Principal Investigator — UBC/VCHA/VGH
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada